CLINICAL TRIAL: NCT06879210
Title: Application of Artificial Intelligence to Construct Whole-person Precise Smart Medicine and Precise Health Care Program in Patients With Myasthenia Gravis
Brief Title: Application of Artificial Intelligence in Precision Medicine and Healthcare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Ting Yeh (Other)
Responsible Party: Sponsor-Investigator, Yi Ting Yeh, Principal Investigator, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20221210R
Record Dates: First submitted 2024-08-10; First posted 2025-03-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; AI
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disease Group (Other): In this study, patients with myasthenia gravis will be used as an example. After the patients use this disease inquiry platform, researchers will conduct interviews with them to understand their experiences and feedback.
  Interventions: Device: Mobile device.(phone)

INTERVENTIONS:
Device: Mobile device.(phone) — Develop a mobile device [Disease Assistance Consultation] to help patients promptly understand their disease and how to care for it. After a 4-week trial period, conduct interviews with participants to determine whether using the mobile device can increase participants' knowledge and improve the quality of healthcare.

SUMMARY:
This study aims to propose an intelligent health robot that utilizes remote intelligent robots to assist patients with disease-related issues, enabling them to address their problems promptly.

DETAILED DESCRIPTION:
Utilizing an information architecture system, a voice-based artificial intelligence program will be developed. The symptoms of major diseases and related knowledge will be input into this system to construct a dedicated disease platform. This platform will allow patients to remotely access it, enabling them to promptly understand and address disease-related issues, thereby improving convenience for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with myasthenia gravis by a physician.
2. Age 20 years and above.
3. Able to use a smartphone.

Exclusion Criteria:

1. Individuals not diagnosed with myasthenia gravis.
2. Individuals who do not use smartphones or tablets.
3. Individuals who withdraw from the group midway.
4. Individuals unwilling to participate in interviews.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Can the use of a mobile device [Disease Assistance Consultation] enhance the understanding of disease care and increase knowledge related to diseases in traditional Chinese medicine? | 4 weeks
  Each patient will be followed up after using the application system for 4 weeks. Each patient will be interviewed for 20 minutes, and the data will be compiled and written later.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Ting Yeh, New Taipei City, Tamsui District, Taiwan